CLINICAL TRIAL: NCT06578169
Title: Initiation of Exogenous Female Sex Hormones and Airway Responsiveness to Methacholine - A Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Erik Soren Halvard Hansen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-23029543
Record Dates: First submitted 2024-08-13; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hormonal Therapy Agent — Women initiating either Hormonal Contraceptives or Hormone replacement therapy in menopause

SUMMARY:
The project aims to investigate the effect of female sex hormone treatment (both contraceptive treatment and hormone therapy during menopause) on bronchial hyperreactivity in adult women. The study is a prospective cohort study involving 300 women, examining airway responsiveness before and after the initiation of hormone treatment, whether as hormone therapy in menopause or contraceptive treatment. Participants will be recruited from general practitioners in the Capital Region of Denmark. Lung function, bronchial hyperreactivity, airway inflammation, and body composition will be assessed before and after hormone treatment. Blood samples will also be collected and stored for later analysis of inflammation markers. The study will include women aged 18 to 75 who are about to begin hormone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 75 years
* Planning to initiate HRT/HC within next 30 days

Exclusion Criteria:

* Gynecological, endocrinological or other disease affecting the ovarian cycle
* FEV1 < 60% of expected or < 1.5L
* Current hormonal medication
* Pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of this study will be women aged 18 to 75 years who for any reason are about to initiate HRT/HC. Further, patients must not be on any hormonal treatment at the time of initiation of hormones and must not have any gynecological or endocrinological disorder which is known to affect the ovarian cycle.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Airway responsiveness to methacholine | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
  Airway responsiveness to methacholine challenge before and after initiation of HC/HRT treatment reported as a dose-response-ratio defined as change in %FEV1 per μmol

SECONDARY OUTCOMES:
Changes in lung function measured as forced expiratory volume in first second (FEV1), forced vital capacity (FVC), | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Change from baseline as measured by airway oscillometry (AOS) | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Changes in airway inflammation measured as FeNO | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Changes in blood alarmins such as blood eosinophils, interleukin 4 (IL-4), IL-5, IL-6, IL-8, IL-10, IL-13, IL-17, IL-23, IL-33, TSLP, IL-1 and Tumor Necrosis Factor alfa (TNF-alfa) | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Medical Research Council Dyspnea Scale (MRC) will be used to evaluate subjective dyspnea. MRC will be evaluated by medical interview. | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Changes in allergy measured as skin prick test (SPT) to common inhaled allergens | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Changes in body composition - fat distribution | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Changes in body composition measured as fat percent | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Changes in body composition measured as fat mass (kg) | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation
Baseline Dyspnea Index (BDI) will be used to evaluate subjective dyspnea. Will be evaluated by medical interview. | 30 to 14 days before initiation of HC/HRT and 7-14 days and 42-56 days following initiation

IPD SHARING:
Plan to Share IPD: Undecided